CLINICAL TRIAL: NCT04104412
Title: The Safety/Efficacy Clinical Study of Human Umbilical Cord Mesenchymal Stem Cells Therapy for Patients With Lumbar Discogenic Pain
Brief Title: The Safety/Efficacy Study of Human Umbilical Cord Mesenchymal Stem Cells Therapy (19#iSCLife®-LDP) for Lumbar Discogenic Pain
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sclnow Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCLnow-XW-01
Record Dates: First submitted 2019-09-02; First posted 2019-09-26 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Lumbar Discogenic Pain
Keywords: lumbar discogenic pain; mesenchymal stem cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group A （with mesenchymal stem cell intervention） (Experimental): observe the effectiveness and safety of patients by injecting human umbilical cord mesenchymal stem cells(2*10^7/ml normal saline) and Low temperature plasma vaporization ablation
  Interventions: Biological: human umbilical cord mesenchymal stem cell
- control group B (No Intervention): observe the effectiveness and safety of patients by injecting normal saline and Low temperature plasma vaporization ablation

INTERVENTIONS:
Biological: human umbilical cord mesenchymal stem cell — 2*10^7
  Arms: treatment group A （with mesenchymal stem cell intervention）

SUMMARY:
This experimental use umbilical cord mesenchymal stem cells in treatment of the early stage of lumbar discogenic pain (endogenous pain of the disc) to evaluate its safety and efficacy.

This experimental is mainly aimed at over 18years old people, regardless of gender, with refractory and persistent back pain for more than 6 months.

The efficacy and safety of mesenchymal stem cells (MSCS) were evaluated by low-temperature plasma ablation and intravertebral disc injection, which were divided into treatment group and control group.

DETAILED DESCRIPTION:
This experimental use umbilical cord mesenchymal stem cells in treatment of the early stage of lumbar discogenic pain (endogenous pain of the disc) to evaluate its safety and efficacy.

This experimental is mainly aimed at over 18years old people, regardless of gender, with refractory and persistent back pain for more than 6 months.

The straight leg elevation test was 70 degrees negative. Magnetic Resonance Imaging (MRI) of the lumbar spine showed herniated disc < 6 mm, no obvious compression of spinal cord and nerve roots. T2-weighted mri of the lumbar spine showed decreased single/multisegment signal in the intervertebral disc (black disc sign) or High intensity zone (HIZ) in the posterior part of the intervertebral disc annulus. The clinical signs of nerve localization were consistent with MRI changes.

The efficacy and safety of mesenchymal stem cells (MSCS) were evaluated by low-temperature plasma ablation and intravertebral disc injection, which were divided into treatment group and control group.

The safety evaluation including:physical examination, vital signs, routine hematuria and faeces, liver and kidney function, blood lipids, electrolytes, coagulation, rapid virus detection, tumor markers, electrocardiogram and adverse reaction records at the 3, 6, 12 and 24 weeks before and after treatment.

The prime efficacy evaluation is VAS( visual analogue scale) at the 3, 6, 12 and 24 weeks before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. age over 18
2. refractory and persistent lumbago pain for more than 6 months, with/without radiation pain in lower limbs, and poor conservative treatment effect;
3. the straight leg elevation test was 70 degrees negative;
4. MRI of lumbar spine showed herniated disc < 6 mm, no obvious compression of spinal cord and nerve roots; T2-weighted mri of the lumbar spine showed decreased single/multi-segment signal (black disc sign) or High signal zone (HIZ) in the posterior part of the intervertebral disc annulus.
5. clinical signs of nerve localization were consistent with MRI changes;
6. subject gives informed consent and signs informed consent.

Exclusion Criteria:

1. coagulation dysfunction or anticoagulant therapy;
2. intervertebral space infection, puncture site infection or systemic infection;
3. lumbago pain of non-spinal origin, such as sacroiliac joint origin pain;
4. patients who have had open surgery or other disc treatments;
5. imaging examination suggested disc prolapse, prolapse, spinal canal bone stenosis, etc.;
6. patients with vital organ system dysfunction and tumor lumbar vertebra metastasis;
7. subjects with high tumor markers (AFP/CEA/CA199/CA125);
8. the subject is pregnant or breastfeeding;
9. subjects also receive other treatments that may affect the efficacy and safety of stem cells;
10. failing to control alcohol and other substance abuse during the 6 months prior to enrollment and enrollment period;
11. the subjects suffer from mental illness, or lack of understanding, communication and cooperation, and cannot be guaranteed to follow the study protocol;

Subjects who are not willing to sign informed consent and are participating in other clinical trials or have participated in other clinical trials within 3 months;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Estimated)
Dates: Start 2019-08-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Validity evaluation by detection the change of the VAS pain score relief rate for Lumbar disc pain of participants in different time point and compare with the VAS pain score before treatment | 24 weeks
  Recording the VAS scores at 3, 6, 12 and 24 weeks after the operation and compare with the VAS score before the operation.
  Pain relief rate =(VAS before treatment - VAS after treatment)/VAS before treatment ×100%.
  VAS scale Use a line with 10 centimeters long as a point between 1 and 10
  0 points, no pain, no pain sensation;
  1-3 points, mild pain, no effect
  4-6 points, moderate pain, affecting work but not life;
  7-10 points, severe pain, severe pain, affect work and life.
  Efficacy evaluation: more than 75% is the basic remission; 50%-75% is effective; 25%-50% effective; Less than 25% is invalid.
  e.g. the VAS score before the operation is 8, the score in the third week after operation is 6, the pain relief rate is (8-6)/8x 100%=14.3% the VAS score before the operation is 8, the score in the sixth week after operation is 3, the pain relief rate is (8-3)/8x 100%=62.5%

SECONDARY OUTCOMES:
Observe treatment | 24weeks
  Secondary measures were assessed at 3, 6, 12 and 24 weeks before and after treatment, including:
  Subjective indicators:
  ODI(The Oswestry Disability Index) score:
  0%-20%: Minimal disability: This group can cope with most living activities. Don't need treatment.
  20%-40% Moderate disability: This group experiences more pain and problems with sitting, lifting, and standing. Personal care, sexual activity, and sleeping are not grossly affected, and the back condition can usually be managed by conservative means.
  40%-60%: Severe disability: Pain remains the main problem in this group of patients, but travel, personal care, social life, sexual activity, and sleep are also affected.
  60%-80%: Crippled: Back pain impinges on all aspects of these patients' lives-both at home and at work-and positive intervention is required.
  80%-100%: These patients are either bed-bound or exaggerating their symptoms. Need evaluated by careful observation of the patient during medical examination.
Safety evaluation by detecting adverse events and serious adverse events | 24 weeks
  Observe for any adverse reactions, including fever, pain, or bleeding to evaluate the changes of safety indexes at the 3、6、12、24weeks after treatment.
Safety evaluation by detecting Activated partial thromboplastin time (APTT) | 24 weeks
  Being the Activated partial thromboplastin time (APTT) test for the patients to examine the changes of safety indexes at the 3、6、12、24 weeks after treatment.
  time of 25-37 seconds. Abnormalities over 10 seconds should be compared with normal controls.
Safety evaluation by detecting Prothrombin time (PT) | 24 weeks
  Being the Prothrombin time (PT) test for the patients to examine the changes of safety indexes at the 3、6、12、24 weeks after treatment.
  time of 11-14 seconds. Abnormalities over 3 seconds in comparison with normal controls are required. Activity: 80-120% INR: 0.8-1.2
Safety evaluation by detecting Fibrinogen | 24 weeks
  Fibrinogen test for the patients to examine the changes of safety indexes at the 3、6、12、24 weeks after treatment.
  The Fibrinogen should in 2-4g/L
Safety evaluation by detecting Thrombin time (TT) | 24 weeks
  Thrombin time (TT) test for the patients to examine the changes of safety indexes at the 3、6、12、24 weeks after treatment.
  the time of 12-16 seconds, TT need to be abnormal for more than 3 seconds compared with normal controls

CONTACTS AND LOCATIONS:
Overall Officials: Yuanzhang Tang, Doctor, Study Director — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No